CLINICAL TRIAL: NCT00322413
Title: Efficacy and Safety of Epoetin Omega in Patients Undergoing Regular Dialysis. Part II: Comparative Trial Versus Epoetin Alfa
Brief Title: Comparison of Epoetin Alfa and Epoetin Omega in Anemic Dialysis Patients:Results of Efficacy Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: General Hospital Sveti Duh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Epo-Comp-00-01
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2006-05

CONDITIONS: End Stage Renal Disease; Renal Anemia; Regular Dialysis Treatment
Keywords: Epoetin alfa; Epoetin omega; Comparative efficacy trial; Renal anemia
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Erythropoietin

INTERVENTIONS:
Drug: Epoetin

SUMMARY:
The two epoetins, Epoetin alfa, a well established drug to treat renal anemia and Epoetin Omega, that differs from Epoetin alfa in the sugar moiety of the molecule were compared in regard of efficacy and safety to treat end stage renal disease anemia. Study hypothesis was that Epoetin Omega is non-inferior to Epoetin alfa in correcting renal anemia in dialysis patients. A 12-weeks randomized comparative efficacy study was performed including 77 end stage renal disease patients (epoetin omega:n=39, epoetin alfa: n=38). In the intent-to-treat analysis, average weekly difference in hemoglobin versus baseline value was higher in omega-treated patients: 1.94+-0.81 vs. 1.23+-0.62 g/dl. The unadjusted and adjusted omega-alfa differences were 0.71 g/dl (95%CI 0.38 to 1.04; p<0.001) and 0.78 g/dl (0.49 to 1.08;p<0.001), respectively. Average weekly epoetin dose was lower in the omega group: 87+-25 vs. 108+-21 IU/kg. The unadjusted and adjusted omega-alfa differences were -21IU/kg (-32 to -11; p<0.001) and -24IU/kg (-35 to -13; p<0.001), respectively. Epoetins were comparably well tolerated. In dialysis patients, subcutaneous epoetin omega apparently provides a greater anti-anemic effect per administered dose (IU) than epoetin alfa.

DETAILED DESCRIPTION:
The two epoetins, Epoetin alfa, a well established drug to treat renal anemia and Epoetin Omega, that differs from Epoetin alfa in the sugar moiety of the molecule were compared in regard of efficacy and safety to treat end stage renal disease anemia. Study hypothesis was that Epoetin Omega is non-inferior to Epoetin alfa in correcting renal anemia in dialysis patients. A 12-weeks randomized comparative efficacy study was performed including 77 end stage renal disease patients (epoetin omega:n=39, epoetin alfa: n=38). All patients were anemic (Hemoglobin < 90 g/L), treated by regular hemodialysis and without signs of bleeding, hemolysis, inflammation or history of major surgery.Treatment was started with 50 IU/kg body weight subcutaneously per week and thereafter adjusted according to the hemoglobin response. In the intent-to-treat analysis, average weekly difference in hemoglobin versus baseline value was higher in omega-treated patients: 1.94+-0.81 vs. 1.23+-0.62 g/dl. The unadjusted and adjusted omega-alfa differences were 0.71 g/dl (95%CI 0.38 to 1.04; p<0.001) and 0.78 g/dl (0.49 to 1.08;p<0.001), respectively. Average weekly epoetin dose was lower in the omega group: 87+-25 vs. 108+-21 IU/kg. The unadjusted and adjusted omega-alfa differences were -21IU/kg (-32 to -11; p<0.001) and -24IU/kg (-35 to -13; p<0.001), respectively. Epoetins were comparably well tolerated. In dialysis patients, subcutaneous epoetin omega apparently provides a greater anti-anemic effect per administered dose (IU) than epoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease
* Regular dialysis treatment
* Renal anemia (hemoglobin<9.0 g/dl)
* Age > 18 years
* Adequate iron stores (TIBC saturation > 20%, ferritin >200)

Exclusion Criteria:

* Signs of bleeding
* Major surgery in previous 60 days
* Hemolysis
* Other causes of anemia
* Cancer
* Inflammatory diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1997-01; Study Completion 1997-04

PRIMARY OUTCOMES:
Hemoglobin level

SECONDARY OUTCOMES:
Average weekly epoetin dose
Time to achieve hemoglobin level of 10 g/dl

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Milutinovic, M.D., Ph.D., Principal Investigator — Department of Nephrology and Dialysis, General Hospital Sveti Duh, Zagreb, Croatia
Locations (1):
- Department of Nephrology and Dialysis, General Hospital Sveti Duh, Zagreb, Croatia

REFERENCES:
- [Result] Milutinovic S, Trkulja V. Reduced responsiveness to epoetin at re-exposure after prolonged epoetin-free period in anemic hemodialysis patients with end-stage renal disease. Croat Med J. 2006 Jun;47(3):424-32. PMID 16758521
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280